CLINICAL TRIAL: NCT07228195
Title: SGLT2i Therapy in Islet Transplantation (SIT)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2025-34226
Record Dates: First submitted 2025-10-17; First posted 2025-11-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Partial Islet Function; TPIAT; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — empagliflozin; Tablets

STUDY DESIGN:
Intervention Model Description: randomized, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- No Medication x 3 months, then 25 mg Empagliflozin x 3 months (No Intervention)
- Empagliflozin 10 mg x 3 months, then 25 mg Empagliflozin x 3 months (Active Comparator)
  Interventions: Drug: Empagliflozin 10 MG Oral Tablet [Jardiance]
- Empagliflozin 25 mg x 6 months (Active Comparator)
  Interventions: Drug: Empagliflozin 25 MG Oral Tablet

INTERVENTIONS:
Drug: Empagliflozin 25 MG Oral Tablet — Empagliflozin, which is sold under the name of Jardiance, is FDA approved for patients 10 years of age and older to improve glycemic control in type 2 diabetes.
  Arms: Empagliflozin 25 mg x 6 months
Drug: Empagliflozin 10 MG Oral Tablet [Jardiance] — Empagliflozin, which is sold under the name of Jardiance, is FDA approved for patients 10 years of age and older to improve glycemic control in type 2 diabetes.
  Arms: Empagliflozin 10 mg x 3 months, then 25 mg Empagliflozin x 3 months

SUMMARY:
This pilot clinical trial is designed to gather preliminary data on the efficacy and safety of empagliflozin, a diabetes drug in the sodium-glucose cotransporter 2 inhibitor (SGLT2i) class, in islet autotransplant recipients who have partial islet function.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old;
* >1 year after TPIAT date at enrollment;
* Partial islet function defined as stimulated C-peptide ≥0.6 ng/mL at screening/baseline visit, AND either (1) on insulin at ≤0.25 unit/kg/day OR (2) not on insulin but HbA1c >6.5%;
* Stable diabetes management defined by stable on pump or multiple daily injections (MDI) for at least 8 weeks and <25% change in insulin dosing over prior 8 weeks.
* Willing to manage diabetes medication management/dose adjustments for the duration of the study with study team MD
* Willing to wear continuous glucose monitor for diabetes management (currently standard of care for TPIAT diabetes)
* Willing to record insulin doses for 14 day intervals x 3 study visits.
* Willing and able to come to the UMN Clinical Research Unit for 3 study visits, approximately 3 months apart
* No prescribed medications other than insulin to treat diabetes in the past 4 weeks.

Exclusion Criteria:

* HbA1c >9%; on any non-insulin antihyperglycemic medication;
* History of diabetic ketoacidosis (DKA) in the past 1 year;
* Unable to drink Boost HP due to true milk protein allergy;
* Underweight (BMI <18.5 kg/m2) [contraindicated by possible weight loss with SGLT2 inhibitors];
* Renal failure defined by glomerular filtration rate <30 mL/min/m2;
* Recurrent dehydration necessitating ED/hospital visits; one time/ rare hospital visits due to intercurrent illness are not exclusionary but repeated dehydration from a chronic condition will be exclusionary.
* Expected to need systemic corticosteroids at >25 mg/day hydrocortisone equivalent over the 6-month study interval;
* Known allergy to empagliflozin;
* Currently pregnant or plan to become pregnant in the next 6 months (for females), or currently breastfeeding;
* Unwillingness to consent or return for study visits;
* Non-English speaking.
* Any other medical contraindication to treatment or study participation in the opinion of the investigator that would impact either patient's safety or their ability to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Time In Range (TIR) 70- 180 mg/dL | Month 3
  the primary comparison is between three treatment arms (control, empagliflozin 10 mg, and empagliflozin 25 mg) at 3 months on treatment

SECONDARY OUTCOMES:
Time in Tight Range (TITR) 70-140 mg/dL | Month 3
  from 14 days of home monitoring
Time in Tight Range (TITR) 70-140 mg/dL | Month 6
  from 14 days of home monitoring
Time in hypoglycemia <70 mg/dL | Month 3
  from 14 days of home monitoring
Time in hypoglycemia <70 mg/dL | Month 6
  from 14 days of home monitoring
Time in hypoglycemia <54 mg/dL | Month 3
  from 14 days of home monitoring
Time in hypoglycemia <54 mg/dL | Month 6
  from 14 days of home monitoring
Time in hyperglycemia >180 mg/dL | Month 3
  from 14 days of home monitoring
Time in hyperglycemia >180 mg/dL | Month 6
  from 14 days of home monitoring
Area under the curve 2 hour glucose from MMTT | Month 3
Area under the curve 2 hour glucose from MMTT | Month 6
Hemoglobin A1c level | Month 3
Hemoglobin A1c level | Month 6
Proinsulin | Month 3
  C-peptide ratios during MMTT at fasting and +90 minutes (beta-cell ER stress marker)
Proinsulin | Month 6
  C-peptide ratios during MMTT at fasting and +90 minutes (beta-cell ER stress marker)
Proportion of patients with ketones >=1.5 | Month 3
  Routine home serum ketone testing
Proportion of patients with ketones >=1.5 | Month 6
  Routine home serum ketone testing
ED/ hospital visits for diabetic ketoacidosis (DKA) | Month 3
  number of visits
ED/ hospital visits for diabetic ketoacidosis (DKA) | Month 6
  number of visits
Occurrence of urinary or genital tract infection | Month 3
Occurrence of urinary or genital tract infection | Month 6
Weight change | Month 3
  % weight loss or weight gain
Weight change | Month 6
  % weight loss or weight gain
Diabetes distress | Month 3
  Diabetes Distress Score; Each item is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem."
Diabetes distress | Month 6
  Diabetes Distress Score; Each item is rated on a 6-point scale from (1) "not a problem" to (6) "a very significant problem."

CONTACTS AND LOCATIONS:
Overall Officials: Melena Bellin, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No